CLINICAL TRIAL: NCT06213805
Title: Efficacy and Safety of Minimally Invasive Micro-Sclerostomy (MIMS) in Glaucoma Surgery
Acronym: MIMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Privé de la Baie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A02193-42
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally invasive microsclerostomy (Experimental)
  Interventions: Procedure: Minimally invasive microsclerostomy

INTERVENTIONS:
Procedure: Minimally invasive microsclerostomy — MIMS is a filtering glaucoma surgery, which consists of creating a sclero-corneal drainage channel, to allow the flow of aqueous humor and therefore the reduction of intraocular pressure.
  This surgery is extremely quick, lasting 3 to 5 minutes, according to recent MIMS studies, in contrast to the duration of a trabeculectomy, the classic glaucoma surgery, which varies between 20 and 60 minutes.

SUMMARY:
The main objective is to evaluate the effectiveness of MIMS in patients with an indication for glaucoma surgery, compared to traditional surgery. The secondary objective is to assess safety. The investigating ophthalmologist will follow the patients and collect clinical data in order to identify the benefits and complications of MIMS. Patients are expected to experience fewer complications compared to traditional glaucoma surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old who agree to participate in the study having signed informed consent
* Primary open-angle glaucoma, pseudoexfoliative glaucoma or pigmentary glaucoma with indication for glaucoma surgery (defined as uncontrolled intraocular pressure or worsening of visual fields, despite maximum tolerated medical therapy) and open iridocorneal angle ( trabecular meshwork visible on gonioscopy, Shaffer classification grade 3-4) and healthy and mobile conjunctiva (without scars or adhesions).
* Chronic angle closure glaucoma with indication for combined glaucoma and cataract surgery

Exclusion Criteria:

* Presence of other ophthalmological pathologies (except cataract)
* History of intraocular surgery (unless cataract surgery), history of trauma, or conjunctival scarring in the quadrant planned for surgery
* Visual acuity lower than "counts fingers" ", closure of the iridocorneal angle (and angle-closure glaucoma unless associated cataract surgery), neovascular glaucoma or neovascularization of the iris, pachymetry < 490 μm or > 620 μm.
* Presence of severe systemic pathologies, pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Measurement of intraocular pressure by tonometry | day 0, day 7, day 14, day 30, month 6, month 9 and month 12 after surgery
  Measure in millimeters of mercury (mmHg)

SECONDARY OUTCOMES:
visual quality of life VFQ-25, | month 1, month 3, month 12 after surgery
  25 questions about visual quality of life with Likert scale (1-5 and 1-6)
Optical Coherence Tomography | month 3, month 12
  high-resolution images of the retina and anterior segment
Visual field test | month 3, month 12
  Measure of visual field in degree (°)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Miguel, MD, Principal Investigator — Hôpital Privé de la Baie
Locations (3):
- France (3):
  - Hôpital Privé de la Baie, Avranches
  - Clinique Thiers, Bordeaux
  - Fondation Rothschild, Paris

IPD SHARING:
Plan to Share IPD: No